CLINICAL TRIAL: NCT00496730
Title: A Multicenter, Randomized, Open Label Study to Evaluate the Lipid Lowering Efficacy and Safety of Vytorin® 10/20 vs. Atorvastatin 10mg in Hypercholesterolemia Patients With Metabolic Syndrome in Korea
Brief Title: A Multicenter, Randomized, Open Label Study to Evaluate the Lipid Lowering Efficacy and Safety of Vytorin® 10/20 vs. Atorvastatin 10mg in Hypercholesterolemia Patients With Metabolic Syndrome in Korea (0653A-129)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0653A-129; MK0653A-129; 2007_017
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
Keywords: Metabolic Disorder
MeSH Terms: conditions — Hypercholesterolemia; Metabolic Diseases | interventions — Ezetimibe, Simvastatin Drug Combination; Atorvastatin

ARMS (2):
- Vytorin® (Experimental): simvastatin (+) ezetimibe 10/20 mg (Vytorin®) ; tablet, once daily, 8 Weeks
  Interventions: Drug: simvastatin (+) ezetimibe
- atorvastatin (Active Comparator): atorvastatin 10 mg; tablet, once daily, 8 Weeks
  Interventions: Drug: Comparator: atorvastatin

INTERVENTIONS:
Drug: simvastatin (+) ezetimibe — simvastatin (+) ezetimibe 10/20 mg ; tablet, once daily, 8 Weeks
  Other Names: MK0653A; Vytorin®
  Arms: Vytorin®
Drug: Comparator: atorvastatin — atorvastatin 10 mg; tablet, once daily, 8 Weeks
  Other Names: Lipitor®
  Arms: atorvastatin

SUMMARY:
Prevalence of metabolic syndrome in korea is increasing. There is no clinical trial targeting on such increasing populations like metabolic syndrome patients with Vytorin® in korea. Therefore this trial will help evaluate the lipid lowering effect of Vytorin® in asian population with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of the metabolic syndrome according to 2005 American Heart Association/National Heart, Lung and Blood Institute (AHA/NHLBI) scientific statement
* No history of diabetes and 100 <=LDL-C <=250 mg/dl

Exclusion Criteria:

* Myocardial Infarction, coronary artery bypass surgery, or angioplasty within 3 months
* Congestive heart failure defined by New York Heart Association (NYHA) class III or IV
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins
* Uncontrolled hypertension
* Unstable angina

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between June 2007 and May 2008.
Pre-assignment Details: Patients who have Metabolic syndrome and Hypercholesterolemia had 4 weeks wash-out period were enrolled in this study. The eligible patients was allocated to one of Vytorin 10/20 mg or Atorvastatin 10 mg group.
Groups:
- Vytorin: simvastatin (+) ezetimibe 10/20 mg (Vytorin®) ; tablet, once daily, 8 Weeks
Period: Overall Study
Arm/Group | Vytorin | Atorvastatin
Started | 130 | 126
Completed | 124 | 121
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vytorin | Atorvastatin | Total
Number analyzed (Participants) | 130 | 126 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.96 (9.42) | 60.26 (9.44) | 59.61 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 79
  Male | 94 | 83 | 177
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.75 (3.59) | 26.45 (3.34) | 26.61 (3.46)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 81.01 (8.47) | 82.11 (8.49) | 81.55 (8.48)
LDL-C (low-Density-Lipoprotein-Cholesterol) [Mean (Standard Deviation); unit: mg/dL] | 159.95 (30.33) | 159.95 (27.34) | 159.95 (28.84)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 130.81 (13.91) | 129.85 (14.51) | 130.34 (14.19)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change of Low Density Lipoprotein-Cholesterol (LDL-C) From Baseline After 8 Weeks.
Time Frame: Baseline and 8 Weeks
Population: All patient treated(APT) approach which included all patients who had baseline measured right before randomization, have taken the study drug more than once after randomization and have one measurement after the initiation of the treatment.
Measure: Mean (Standard Deviation); unit: Percent of Baseline Value
Arm/Group | Vytorin | Atorvastatin
Number analyzed (Participants) | 124 | 121
Percent of Baseline Value | -49.29 (15.22) | -38.05 (12.28)
Statistical Analysis 1: Comparison: Vytorin vs Atorvastatin; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Number of Patients Attaining LDL-C Goal After 8 Weeks Treatment.
Description: Number of Patients Attaining LDL-C Goal After 8 Weeks Treatment.
  LDL-C goal is based on National Cholesterol Education Program (NCEP) III guideline (LDL-C goals and cutpoints for therapeutic life changes and drug Therapy in different risk).
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Number; unit: Participants attaining LDL-C goal
Arm/Group | Vytorin | Atorvastatin
Number analyzed (Participants) | 124 | 121
Participants attaining LDL-C goal | 105 | 93
Statistical Analysis 1: Comparison: Vytorin vs Atorvastatin; Test type: Superiority or Other; p < 0.0001, ANCOVA

3. Other Pre Specified Outcome: Change in Lower Density Lipoprotein Cholesterol From Baseline After 8 Weeks.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vytorin | Atorvastatin
Number analyzed (Participants) | 124 | 121
mg/dL | 83.52 (33.84) | 98.27 (21.82)
Statistical Analysis 1: Comparison: Vytorin vs Atorvastatin; Test type: Superiority or Other; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Arm/Group | Vytorin | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 1 | 1
Other Adverse Events (participants affected / at risk) | 25 | 29
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Vytorin | Atorvastatin
Hepatic enzyme increased (Investigations) | 0/124 (0) | 1/121 (2)
Death (General disorders) | 1/124 (1) | 0/121 (0)
Pyrexia (General disorders) | 0/124 (0) | 1/121 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Vytorin | Atorvastatin
Hepatic enzyme increased (Investigations) | 2/124 (3) | 3/121 (4)
High Density lipoprotein decreased (Investigations) | 2/124 (2) | 5/121 (5)
Blood Insulin Increased (Investigations) | 2/124 (2) | 0/121 (0)
Blood creatine phosphokinase increased (Investigations) | 1/124 (1) | 0/121 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0/124 (0) | 1/121 (1)
Bood Urea Increased (Investigations) | 0/124 (0) | 1/121 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6/124 (6) | 6/121 (7)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 4/124 (4) | 3/121 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0/124 (0) | 1/121 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2/124 (2) | 1/121 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2/124 (2) | 1/121 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1/124 (1) | 0/121 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1/124 (1) | 0/121 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2/124 (2) | 3/121 (3)
Abdominal pain lower (Gastrointestinal disorders) | 1/124 (1) | 0/121 (0)
Ascites (Gastrointestinal disorders) | 1/124 (1) | 0/121 (0)
Nausea (Gastrointestinal disorders) | 1/124 (1) | 0/121 (0)
Diarrhoea (Gastrointestinal disorders) | 0/124 (0) | 2/121 (3)
Toothache (Gastrointestinal disorders) | 1/124 (1) | 0/121 (0)
Vomiting (Gastrointestinal disorders) | 0/124 (0) | 1/121 (1)
Headache (Nervous system disorders) | 2/124 (2) | 3/121 (3)
Hypoaesthesia (Nervous system disorders) | 1/124 (1) | 0/121 (0)
Neurological symptom (Nervous system disorders) | 1/124 (1) | 0/121 (0)
Dizziness (Nervous system disorders) | 0/124 (0) | 3/121 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/124 (1) | 0/121 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1/124 (1) | 0/121 (0)
Death (General disorders) | 1/124 (1) | 0/121 (0)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0/124 (0) | 1/121 (1)
Pyrexia (Respiratory, thoracic and mediastinal disorders) | 0/124 (0) | 1/121 (1)
Upper respiratory tract infection (Infections and infestations) | 1/124 (1) | 3/121 (3)
Pneumonia (Infections and infestations) | 0/124 (0) | 1/121 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/124 (1) | 0/121 (0)
Dysuria (Renal and urinary disorders) | 1/124 (1) | 0/121 (0)
Tinnitus (Renal and urinary disorders) | 0/124 (0) | 1/121 (1)
Eye pain (Eye disorders) | 0/124 (0) | 1/121 (1)
Myodesopsia (Eye disorders) | 0/124 (0) | 1/121 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0/124 (0) | 1/121 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0/124 (0) | 1/121 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0/124 (0) | 1/121 (1)
Peripheral coldness (Vascular disorders) | 0/124 (0) | 1/121 (1)
Hypertension (Vascular disorders) | 0/124 (0) | 1/121 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes